CLINICAL TRIAL: NCT01756521
Title: A Multi-center, Randomized, Open-label, Placebo-controlled, 3-way Crossover Study to Investigate the Effect on QT/QTc Interval of Moxifloxacin After a Single Dose in Healthy Male Subjects
Brief Title: A Study Study to Investigate the Effect on QT/QTc Interval of Moxifloxacin After a Single Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea National Enterprise for Clinical Trials (Other); The Catholic University of Korea (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Sang Yu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MOXI036
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: the Effect of Moxifloxacin on QT/QTc Interval
Keywords: QT,; QTc,; electrocardiogram,; moxifloxacin
MeSH Terms: interventions — Moxifloxacin

ARMS (3):
- Moxifloxacin 400mg (Experimental): moxifloxacin 400mg
  Interventions: Drug: Moxifloxacin
- Moxifloxacin 800mg (Experimental): moxifloxacin 800mg
  Interventions: Drug: Moxifloxacin
- Placebo(No treatment) (Placebo Comparator): Only drink water
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate effect of moxifloxacin on QT/QTc interval in healthy male subjects. Moxifloxacin is a positive control drug used in QT study. In this study, moxifloxacin 400mg and 800mg will be used, to get information on effect of moxifloxacin on QT/QTc interval.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate effect of moxifloxacin on QT/QTc interval in healthy male subjects. Moxifloxacin is a positive control drug used in QT study. In this study, moxifloxacin 400mg and 800mg will be used, (therapeutic and supratherapeutic doses) to get information on effect of moxifloxacin on QT/QTc interval in healthy Korean male subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subject aged 20 to 40 at screening
* subjects who have weight over 50 kg with ideal body weight range of +- 20%
* subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have acute illness within 28 days of investigational drug administration
* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* subjects who have determined not eligible by screening test (medical history, physical examination, 12-lead ECG, laboratory test, etc) within 28 days of study start
* clinically significant allergic disease (except for mild allergic rhinitis)
* systolic blood pressure>= 140 mmHg, diastolic blood pressure >= 90 mmHg, heart rate > 100 bpm or < 50 bpm
* result of 12-lead electrocardiogram includes :

  * QTcF > 450 msec
  * PR interval > 200 msec or <110msec
  * Evidence of second- or third-degree atrioventricular (AV) block
  * Pathologic Q waves (defined as Q-wave > 40 msec or depth > 0.5 millivolt
  * Evidence of ventricular pre-excitation, left bundle branch block (LBBB), right bundle branch block (RBBB)
  * Intraventricular conduction delay with QRS > 120 msec
* risk of Torsade de pointes such as long QT syndrome, family history of sudden death, heart failure, hypokalemia
* Subjects considered unsuitable for inclusion by the investigator

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
QTc (QTcF, QTcB, QTcI) | Day1 and Day2 of each periods(3 periods)
  QTc (QTcF, QTcB, QTcI)
  * QTcF (Fridericia-corrected QTc)
  * QTcB (Bazett-corrected QTc)
  * QTcI (Individual-corrected QTc)
  QTc change: the largest time-matched, baseline-adjusted least squares mean difference time-matched, baseline-adjusted least squares mean difference

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Ph.D., Principal Investigator — Seoul National University Hospital and College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- See also: webpage of clinical trial center of Seoul National University Hospital — http://ctc.snuh.org